CLINICAL TRIAL: NCT05749107
Title: In-depth Characterization of Atriogenic Secondary Tricuspid Regurgitation Due to Atrial Fibrillation. Prevalence, Mechanisms, Advanced Quantification of Regurgitation Severity, and Relative Impact of Sinus Rhythm Restoration on the 3D Remodeling of Right Heart Chambers and Tricuspid Valve Apparatus
Brief Title: In-depth Characterization of Atriogenic Secondary Tricuspid Regurgitation Due to Atrial Fibrillation
Acronym: ASTRA
Status: Recruiting | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Collaborators: Ministry of Health, Italy (Other Government)
Responsible Party: Sponsor
Other Study IDs: 09M202
Record Dates: First submitted 2023-02-18; First posted 2023-03-01 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Heart Valve Incompetence; Atrial Fibrillation, Persistent
Keywords: Functional tricuspid regurgitation; Three-dimensional echocardiography; Doppler echocardiography; Right ventricular function; Atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Biospecimen Retention: Samples Without DNA — Serum and plasma specimen for proteomic and miRNA analyses
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Atrial secondary tricuspid regurgitation: Patients with persistent/permanent atrial fibrillation and any degree of isolated tricuspid regurgitation
  Interventions: Diagnostic Test: Echocardiography; Combination Product: Proteomic analyses

INTERVENTIONS:
Diagnostic Test: Echocardiography — Identify AF patients at risk of developing moderate/severe STR and those who will benefit from restoring the normal sinus rhythm
Combination Product: Proteomic analyses — To identify the mechanisms leading to moderate/severe STR during AF.

SUMMARY:
1050 patients with persistent/permanent atrial fibrillation (AF) will be studied using conventional and advanced (three-dimensional and deformation imaging) echocardiography. Patients with moderate/severe isolated secondary tricuspid regurgitation (STR) will undergo blood tests to assess their proteomic profile and cardiac CT to measure the tricuspid annulus geometry. The project will aim to 1. assess the prevalence of moderate/severe isolated STR in patients with AF; 2. identify the mechanisms associated with the development of moderate-severe STR in patients with AF; 3. identify the proteomic profile associated with significant growth of tricuspid valve leaflets as a mechanism to protect patients with AF from the development of moderate/severe STR; 4. evaluate the effects of the restoration of sinus rhythm on the severity of STR and the remodeling of the right heart cardiac structures (i.e. right ventricle, right atrium, and tricuspid valve apparatus).

ELIGIBILITY:
Inclusion Criteria:

* age> 18 years
* persistent/permanent atrial fibrillation
* good acoustic apical window
* left ventricular ejection fraction > 50%
* pulmonary artery systolic pressure< 50 mm Hg
* no more than mild mitral or aortic valve disease
* ability to attend clinical and echocardiographic follow-ups
* signature of the study informed consent

Exclusion Criteria:

* pregnancy
* implanted pace-maker or ICD
* previous heart valve surgery or transcatheter treatment
* previous heart transplant
* organic tricuspid regurgitation

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing echocardiography stud because of persistent/permanent atrial fibrillation
Sampling Method: Non-Probability Sample
Enrollment: 1050 (Estimated)
Dates: Start 2022-12-02 (Actual); Primary Completion 2024-12-02 (Estimated); Study Completion 2025-11-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of either moderate or severe functional tricuspid regurgitation | 1 year
  To assess the prevalence of moderate or severe atriogenic secondary tricuspid regurgitation (STR) in patients with persistent/permanent atrial fibrillation (AF), and to develop valve-specific metrics and parameters to assess STR severity by echocardiography.
To identify the mechanisms leading to moderate/severe STR during AF. | 3 years
  STR severity varies among patients with persistent/permanent AF and comparable RV and RA remodeling. The role of RV and RA size, shape, and function on the extent of tricuspid annulus dilation and dysfunction remains to be clarified.
  Moreover, it is unknown whether the leaflets of the tricuspid valve can adapt to the stretch exerted on them by the progressive dilation of the tricuspid annulus. The contribution of leaflet adaptation to the pathophysiology of STR and its molecular determinants remains to be clarified
To evaluate the extent of the right heart structure remodeling occurring after the recovery of the sinus rhythm and its effects on STR severity. | 3 years
  Patients undergoing sustained cardioversion to sinus rhythm (both electrical and pharmacological) and/or ablation of AF, will be followed at 1, 3, and 12 months after the procedure by recording electrocardiogram and complete 2D Doppler and 3DE to assess the extent of the remodeling of the RV, the RA, and the tricuspid valve apparatus. Patients with atriogenic moderate/severe STR without clinical indication to either cardioversion or ablation of the AF, and patients with none/mild atriogenic STR will be followed with clinical assessment, and complete 2D, Doppler and 3DE at 6 months and 1 year.
  The severity of STR will be quantified by measuring EROA, regurgitant volume, and regurgitant fraction.

SECONDARY OUTCOMES:
Development of an interpretable predictive model by using and integrating a variety of statistical and artificial intelligence (AI) techniques. | 3 years
  Clinical, echocardiographic, and biomarker parameters that might predict either the development of moderate/severe STR in patients with AF or the likelihood of reduction of STR severity after cardioversion in sinus rhythm will be identified and integrated in an expert system based on fuzzy reasoning.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Istituto Auxologico Italiano, IRCCS, Milan, Select A State
  - IRCCS Ospedale San Raffaele, Milan

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available upon reasonable request
Supporting Information: Study Protocol, ICF
Time Frame: Available now, till the end of the study
Access Criteria: Data will be made available upon reasonable request